CLINICAL TRIAL: NCT05516563
Title: An EDucation and eXercise Intervention (EDX-Ireland) for Gluteal Tendinopathy in an Irish Setting: a Feasibility Randomised Controlled Trial (LEAP-Ireland Trial)
Brief Title: LEAP-Ireland Feasibility Trial of Exercise and Education for Gluteal Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoyalCSILeapIreland
Record Dates: First submitted 2022-07-27; First posted 2022-08-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-05

CONDITIONS: Gluteal Tendinopathy; Trochanteric Bursitis; Greater Trochanteric Pain Syndrome
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: A feasibility randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDucation and eXercise intervention (EDX) (Active Comparator): EDX-Ireland will involve 6 face-to-face education and exercise sessions on a individualised basis with a physiotherapist, delivered over eight weeks. This will be supplemented by a home based exercise programme.
  Interventions: Other: EDucation and eXercise intervention
- Usual Care (No Intervention): Participants will continue to follow what they have done so far for their hip pain, or what their doctor has suggested/prescribed. If a participant is referred to physiotherapy as part of the usual care treatment, waiting time will be recorded.
  Participants will receive a written information leaflet on the pathology of gluteal tendinopathy and general advice on symptom management.

INTERVENTIONS:
Other: EDucation and eXercise intervention — The exercise programme includes 3 key streams:
  1. Low-load isometric abduction
  2. Functional loading
  3. Abductor loading: Graduated abductor loading, designed to improve load tolerance by applying progressively higher loads across the abductor muscles. Daily exercise will be completed three days a week at a 'hard' to 'very hard' level, alternating with three 'light' days and one rest day. The clinic day will constitute one of the 'hard' days.
  Education will be delivered via a 20 minute video which focusses on understanding and managing lateral hip pain ( ie pain associated with gluteal tendinopathy). Education will also be tailored to each patient on attendance with the physiotherapist at the 6 clinic visits
  Arms: EDucation and eXercise intervention (EDX)

SUMMARY:
Gluteal tendinopathy, a degenerative condition of the gluteal tendons, is a common cause of lateral hip pain. It is three times more common in women, affecting up to 25% of those aged over 40 years. Research evidence supporting the most effective interventions remains limited. A 2018 landmark three-arm RCT (LEAP trial) in Australia compared EDucation on load management plus eXercise (EDX) against corticosteroid injection (CSI), and a 'wait-and see' control on pain and global improvement in 205 individuals with gluteal tendinopathy (Mellor et al, 2016; 2018). Results showed superior and significant positive effects in the EDX group, compared with CSI and wait-and-see groups at 8 weeks and 1 year. A total of 14 EDX sessions was provided over 8 weeks in LEAP, but in the public healthcare system in Ireland, typically 5-6 physiotherapy treatments are provided.

Therefore, whilst the LEAP trial demonstrated positive effects for EDX, implementation into clinical practice in Ireland is questionable as 6 or less treatment sessions are typically provided in public and private settings in Ireland (French et al, 2020). This two-arm feasibility RCT aims to evaluate the feasibility of conducting a future RCT of a reduced dose (6 sessions) of a recently proven efficacious physiotherapy treatment of EDucation plus eXercise (EDX-Ireland) to usual care for gluteal tendinopathy in an Irish setting. A Study Within A Trial will evaluate if exercise adherence is improved with use of a smartphone app compared with paper-based diaries.

DETAILED DESCRIPTION:
Study design: A two-arm assessor-blinded feasibility RCT will be conducted, incorporating a Study Within a Trial (SWAT) and embedded qualitative research. The CONSORT statement for pilot and feasibility randomised studies will be followed in the conduct and reporting of this trial.

Participants: Patients with gluteal tendinopathy in Ireland can present to their GP, self-refer to private physiotherapy, or attend secondary care rheumatology clinics. Various recruitment sources will be targetted in this feasibility trial, including: community recruitment, GP practices, sports medicine physicians and secondary care rheumatology or musculoskeletal triage clinics to establish optimal recruitment methods for a full-scale RCT. The following recruitment sources in the greater Dublin area will be notified of the study, provided with study information and a meeting arranged with the trial manager, if they are interested in being a recruitment source.

Procedure: Potential participants will initially be informed of the trial through the recruitment sites (hospitals and GPs), social media or through sports/leisure clubs and organisations. A study invitation letter will be sent out to all recruitment sites. This will also include a participant information sheet providing details of the study, participant eligibility criteria, and clear instructions on how to participate.

If participants indicate a willingness to hear more about the trial, the referral source will provide a leaflet/invitation with contact information of the trial manager and a link to the trial webpage and the Participant Information Leaflet. Interested participants will be initially screened via a phone screening procedure to ensure their eligibility. Those who progress through phone screening, will be invited to schedule an appointment for physical screening with the trial manager.

Once a person has successfully passed physical screening, an appointment will be made for them to attend for a hip MRI by the trial manager. Presence of MRI-confirmed gluteal tendinopathy will deem the person eligible for study inclusion. Participants will be informed that they can withdraw at any stage from the trial.

Participants will be randomised to one of two groups

1. 6 physiotherapy sessions of exercise and education over 8 weeks
2. Usual Care

Experienced registered physiotherapists will deliver the EDX-Ireland intervention. Load management information, exercises and a diary for recording treatment adherence will be provided to the EDX-Ireland group through PhysiApp and Physitrack, Physitrack is an online exercise management system used by physiotherapists for exercise prescription (www.physitrack.com). PhysiApp is the companion platform used by patients to access video-based exercises and education prescribed. As part of the SWAT, the EDX group will be randomly allocated to one of two groups. Both groups will use the PhysiApp for the home exercises but Group A will use the PhysiApp to record their exercise adherence, while Group B will use the paper-based diary format provided by their physiotherapist.

Co-interventions: Participants will be advised not to use other types of treatments, other than the usual care that their referring practitioner has provided, during the 8-week period if possible. Any additional healthcare use will be recorded at both 8-week and 3-month follow-up for cost-effectiveness analysis.

Clinical and Patient Reported Outcomes (PROs) to be collected at baseline, 8 weeks and 3 months are mapped to the LEAP trial and core domains identified by an international consensus group in tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 35-70 years
* Lateral hip pain for at least 3 months, of ≥ 4/10 on an 11-point numeric rating scale on most days of the last 3 months
* Tenderness on palpation of the greater trochanter
* Reproduction of pain on at least one of following diagnostic clinical tests: (FADER test, FADER with Static muscle test (internal rotation) at end of range (FADER-R), FABER test, passive hip Adduction in side lying (ADD) test, adduction with resisted isometric abduction (ADD-R), and single leg stand (SLS) for 30 seconds
* Demonstrated tendon pathology on MRI
* Access to a computer, smartphone or tablet with internet connection

Exclusion Criteria:

* Previous cortisone injection in the region of the lateral hip in the last 12 months
* Physiotherapy (including regular appropriate Pilates) for lateral hip pain in the last 3 months
* Lumbar spine or lower limb surgery in the last 6 months
* Any known advanced hip joint pathology where groin pain is the primary complaint and/or where groin pain is experienced at an average intensity of ≥2 on most days of the week, or Kellgren-Lawrence score of >2 (mild) on X-Ray
* If the following clinical criteria for the diagnosis of hip osteoarthritis (American College Rheumatology) are fulfilled:

  * Self-reported hip pain with either hip internal rotation <15° and hip flexion ≤115° or ≥15° hip internal rotation and pain on hip internal rotation
  * Μorning stiffness ≤ 60 minutes
  * Αge ≥ 50 years
* Hip joint flexion is <90°, bilaterally
* Lumbar radiculopathy or pain in another body location that is greater than the hip pain (NRS)
* Known advanced knee pathology or restricted knee range of motion (must have minimum 90° flexion and full extension, bilaterally)
* Any systemic diseases affecting the muscular or nervous system, and uncontrolled diabetes
* Fibromyalgia
* Use of cane or walking aid
* Malignant tumour (current or in the past 6 months)
* Systemic inflammatory disease
* Any factors that would preclude the participant from having an MRI (e.g. pacemaker, metal implants, pregnancy, or trying to become pregnant, claustrophobia)
* If the participant is involved in any injury claim
* If the participant is unable to commit to an 8-week programme of up to 6 sessions of exercise
* If the participant is unable to write, read or comprehend English
* Unable or unwilling to use technology for exercise prescription and adherence

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 3:1
Enrollment: 65 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Success of different patient recruitment methods (including community recruitment, primary care and secondary care) | Through study completion, an average of 1 year
  Number of participants recruited using different recruitment methods, and the number retained at the 8-week and 3-month time-points will be recorded.
Usual care treatment/recommendations for Gluteal Tendinopathy in Ireland | Through study completion, an average of 1 year
  The constituents of care received from the referral source (GP, orthopedics, rheumatologists, musculoskeletal triage physiotherapists) for Gluteal Tendinopathy in Ireland will be assessed at baseline for all those allocated to the usual care arm
Cost-effectiveness information of Gluteal Tendinopathy in Ireland | Baseline, 8 weeks and 3 months
  Healthcare costs change from baseline, at 8 weeks and 3 months (including pain medication usage, GP visits, investigations, attendance at physiotherapy/other healthcare practitioners or hospital attendance) by trial participants for their hip pain will be recorded.

SECONDARY OUTCOMES:
Pain severity - Numeric Pain Rating scale (NPRS) | baseline, and at 8weeks, and 3months
  Pain severity will be ascertained using a Numeric Pain Rating scale (NPRS) under two conditions of pain on activity/loading and pain in the last week. The NPRS is an 11-point scale with anchors of no pain at 0 and worst pain at 10.
VISA Gluteal (VISA-G) | baseline, and at 8weeks, and 3months
  VISA Gluteal (VISA-G) is a self-reported questionnaire specifically developed to measure disability associated with gluteal tendinopathy.
Patient-Specific Functional Scale (PSFS) | baseline, and at 8weeks, and 3months
  The Patient-Specific Functional Scale (PSFS) is a self-reported, patient-specific measure, designed to assess functional change in patients with musculoskeletal conditions. It has the advantage of being specific to an individual, who is asked to identify three important activities they are unable to perform or are having difficulty with because of their hip problem. They rate the current level of difficulty associated with each activity on an 11- point scale.
Patient Health Questionnaire-9 (PHG-9) | Baseline, 8 weeks and 3 months
  The Patient Health Questionnaire (PHQ-9) is a valid and reliable self-reported questionnaire for measurement of depressive symptoms. It contains nine questions with a score range of 0-27. A score of ≥5 indicates mild depressive symptoms, ≥10 moderate, ≥15 moderately severe and ≥ 20 severe.
The EuroQol 5-D-5L | Baseline, 8 weeks and 3 months
  The EuroQol 5-D-5L is a generic measure of health-related quality of life (HR-QOL). It includes domains of mobility, personal care, usual activities, pain and anxiety/depression that best describe their health status, as well as a single index value for health status.
The Central Sensitisation Inventory (CSI) | Baseline, 8 weeks and 3 months
  The Central Sensitisation Inventory (CSI) is a self-reported screening instrument designed to identify presence of centrally-mediated pain sensitisation. It comprises 25 questions related to symptoms associated with Central Sensitisation. A cut-off score of '40' of '100' yielded good sensitivity (81%).
Global Rating of Change (GROC) | Baseline, 8 weeks and 3 months
  The Global Rating of Change (GROC) is an 11-point ordinal scale which is completed by the patient based on their perceived overall change in their hip condition and allows patients to consider factors that they consider important for their clinical situation. It is anchored by 'very much better' and 'very much worse'.
Pain Catastrophising Scale | Baseline, 8weeks, and 3 months
  The Pain Catastrophising Scale (PCS) is a valid and reliable 13-item self-report measure, which asks about thoughts and feelings associated with pain. It produces a total score, and three subscale scores, which assess rumination, magnification and helplessness.
Pain Self-Efficacy Questionnaire | Baseline, 8 weeks and 3 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a self-reported questionnaire that assesses the confidence that people have in performing activities when they are in pain. It contains 10 items answered on a 7-point Likert scale. It provides clinicians with a quick and easy guide as to how a patient may respond to an activity upgrade or exercise program.
Isometric Hip Abductor Muscle Strength | Baseline, 8 weeks and 3 months
  Isometric Hip Abductor Muscle Strength will be tested in supine using a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- RCSI, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] French HP, Woodley SJ, Fearon A, O'Connor L, Grimaldi A. Physiotherapy management of greater trochanteric pain syndrome (GTPS): an international survey of current physiotherapy practice. Physiotherapy. 2020 Dec;109:111-120. doi: 10.1016/j.physio.2019.05.002. Epub 2019 Jun 2. PMID 31493863
- [Background] Mellor R, Bennell K, Grimaldi A, Nicolson P, Kasza J, Hodges P, Wajswelner H, Vicenzino B. Education plus exercise versus corticosteroid injection use versus a wait and see approach on global outcome and pain from gluteal tendinopathy: prospective, single blinded, randomised clinical trial. BMJ. 2018 May 2;361:k1662. doi: 10.1136/bmj.k1662. PMID 29720374
- [Background] Gundogan UN, Turker RK. Influence of pulmonary circulation on diuretic action of prostaglandin E2. Pharmacology. 1974;11(5):278-86. doi: 10.1159/000136500. No abstract available. PMID 4852446
- [Derived] Almousa S, Vicenzino B, Mellor R, Grimaldi A, Bennett K, Doyle F, McCarthy GM, McDonough SM, Ryan JM, Lynch K, Sorensen J, French HP. An EDucation and eXercise intervention for gluteal tendinopathy in an Irish setting: a protocol for a feasibility randomised clinical trial (LEAP-Ireland RCT). HRB Open Res. 2024 Jun 28;6:76. doi: 10.12688/hrbopenres.13796.2. eCollection 2023. PMID 39045032